CLINICAL TRIAL: NCT07135609
Title: Apitoxin Versus Soft Laser for Management of Aphthous Ulceration
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Omar Elboraey Elbal, Assistant Professor of Oral Medicine, Periodontology, Oral Diagnosis and Oral Radiology Department, Faculty of Dentistry, Tanta, University, Tanta, Egypt, Tanta University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TUCDREC/300424/ Rsabra.
Record Dates: First submitted 2025-08-14; First posted 2025-08-22 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Apitoxin; Bee Venom Therapy; Management; Aphthous Ulceration
MeSH Terms: conditions — Foot-and-Mouth Disease | interventions — Low-Level Light Therapy; Bee Venoms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group Ӏ (Active Comparator): Patients managed by Low-level laser therapy (LLLT).
  Interventions: Device: Low-level laser therapy (LLLT)
- Group II (Experimental): Patients managed with 0.3% Apitoxin Gel.
  Interventions: Drug: Apitoxin

INTERVENTIONS:
Device: Low-level laser therapy (LLLT) — Patients managed by Low-level laser therapy (LLLT).
  Arms: Group Ӏ
Drug: Apitoxin — Patients managed with 0.3% Apitoxin Gel.
  Arms: Group II

SUMMARY:
The current study evaluated the clinical effect and outcome of locally applied bee venom versus low-level laser therapy (LLLT) for the treatment of recurrent aphthous ulceration.

DETAILED DESCRIPTION:
Recurrent aphthous stomatitis (RAS) is a Painful, idiopathic, and recurrent inflammatory ulceration of the oral cavity.

Despite their widespread use, prolonged or frequent application may result in adverse effects such as oral candida. In recent years, low-level laser therapy (LLLT) has gained attention as an alternative treatment for RAS.

Apitoxin has been used traditionally to treat a variety of conditions, such as arthritis, rheumatism, back pain, cancer, and skin diseases.

ELIGIBILITY:
Inclusion Criteria:

* Age from 15 to 40 years old.
* Both sexes.
* No current or history of systemic medical problem.
* Non-smoker.
* Suffering from pain due to recurrent aphthous stomatitis (RAS) ulceration on the oral mucosa with the following characteristics:
* Duration of 2 days or less.
* The diameter ≥ 4mm
* Not been subjected to any treatment modalities for at least four weeks before the beginning of the study.

Exclusion Criteria:

* Presence of other oral mucosal ulcers other than RAS.
* Systemic disease that predisposed them to RAS (e.g., Behçet disease).
* Systemic medical problems.
* Pregnant, lactating, and postmenopausal patients.
* Smoker patients.
* Systemic or topical treatment for RAS less than four weeks before starting the study.
* Any earlier experiences of laser therapy.

Ages: 15 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-04-30 (Actual); Primary Completion 2025-02-02 (Actual); Study Completion 2025-02-02 (Actual)

PRIMARY OUTCOMES:
Ulcer Surface Area | 5 days post-treatment
  Ulcer Surface Area: The main outcome will be the objective measurement of the ulcer surface area. This was evaluated through photographs taken on Day 1 (baseline) and Day 5 (post-treatment).

SECONDARY OUTCOMES:
Pain Sensation | 5 days post-treatment
  Subjective evaluation of pain sensation using the Visual Analog Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). Pain will be assessed on Day 1 (baseline) and Day 5 (post-treatment).
Effectiveness Index (EI) | 5 days post-treatment
  Calculated improvement in pain sensation for each patient based on baseline and post-treatment Visual Analog Scale (VAS). Formula: (VAS baseline - VAS post-treatment) / VAS baseline × 100%

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.